CLINICAL TRIAL: NCT02435121
Title: Phase II, Open Label, Single Arm Study Assessing the Clinical Benefit of SAR125844, Administered as Single Agent by Weekly Intravenous (IV) Infusion, for the Treatment of Patients With Advanced Pretreated Non-Small Cell Lung Cancer (NSCLC) Harboring MET Gene Amplification
Brief Title: A Study Assessing Efficacy and Safety of SAR125844 in NSCLC Patients With MET Amplification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT14205; 2014-005696-93 (EudraCT Number); U1111-1163-1136 (Other: UTN)
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — SAR125844

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR125844 (Experimental): Given intravenously weekly at the dose of 570 mg/m^2 for at least 18 weeks
  Interventions: Drug: SAR125844

INTERVENTIONS:
Drug: SAR125844 — Pharmaceutical form:Concentrate for solution Route of administration: intravenous

SUMMARY:
Primary Objective:

To determine objective response rate (ORR).

Secondary Objectives:

To assess duration of response (DR), progression free survival (PFS) and overall survival (OS).

To evaluate global safety profile. To determine pharmacokinetic profile. To assess clinical utility of fluorescence in situ hybridization (FISH) assay in selection of patients with mesenchymal-epithelial hybridization (MET) gene amplification.

To assess lung cancer symptoms, health-related quality of life and treatment satisfaction.

DETAILED DESCRIPTION:
The duration of the study for 1 patient will include a screening period of up to 3 weeks, a 3-week treatment cycle(s) and a follow-up period. The patients will be treated for 6 cycles in case no response is observed, and treatment may be continued beyond 6 cycles in case of partial response/complete response (PR/CR) or significant clinical benefit until progressive disease, unacceptable toxicity, willingness to stop the study treatment or until study termination by sponsor. After the completion of the study treatment each patient will be followed every 6 weeks until death or the study cut-off date, whichever comes first. For patients who went-off study treatment prior disease progression is documented, date of disease progression and further anticancer treatment will be collected in follow-up visit.

The cut-off date corresponds to the date at which all the treated patients will have 3 post-baseline tumor assessments or will early discontinue whatever the reason. Beyond cut-off date, patient can continue study treatment until disease progression, unacceptable toxicity or patient's refusal, provided clinical benefit is established.

ELIGIBILITY:
Inclusion criteria:

Metastatic non-small-cell lung cancer patients with progressive disease during or after first or second line therapy harboring MET gene amplification and with measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

Exclusion criteria:

Patient less than 18 years old. Eastern Cooperative Oncology Group (ECOG) performance status >2. More than 2 episodes of disease progression under anticancer therapy. Wash out period of less than 3 weeks from prior treatment with chemotherapy, radiotherapy or, surgery or any investigational treatment.

Adequate hematologic, hepatic, renal, coagulation, and metabolic functions. No resolution of any specific toxicities (excluding alopecia) related to any prior anti-cancer therapy to grade ≤1 according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.03.

Pregnant or breast-feeding women. Patient with reproductive potential without method of contraception. Symptomatic brain metastasis. Any clinically significant medical condition other than cancer which could interfere with the safe delivery of study treatment or risk of toxicity.

Known hypersensitivity or any adverse event related to the study drug excipient (Captisol®).

Prior treatment with any MET Tyrosine Kinase Inhibitors (TKIs) or anti-MET antibodies (excluding onartuzumab).

Patients treated with potent CYP3A inhibitor unless it can be discontinued. Patients treated with potent and moderate CYP3A inducers unless it can be discontinued.

Mean QTc interval prolongation >470 msec.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Determination of the objective response rate of SAR125844 as per RECIST 1.1 | every 6 weeks up to 34 months

SECONDARY OUTCOMES:
Progression-free survival rate | up to 34 months
Overall survival rate | up to 34 months
Proportion of patients with adverse events | up to 40 months
Assessment of pharmacokinetic parameters: maximum plasma concentration (Cmax) | up to 3 days
Assessment of pharmacokinetic parameters: area under curve (AUC) | up to 3 days
Assessment of pharmacokinetic parameters: total clearance (CL) | up to 3 days
Assessment of pharmacokinetic parameters: half-life (t1/2) | up to 3 days
Assessment of lung cancer symptoms by Core Quality of Life questionnaire (QLQ-C30) +LC13 | every 3 weeks up to 34 months
Assessment of health-related quality of life by QLQ-C30/LC13 | every 3 weeks up to 34 months
Assessment of treatment satisfaction by Cancer Therapy Satisfaction Questionnaire | every 6 weeks up to 34 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 056001, Edegem, Belgium